CLINICAL TRIAL: NCT03553654
Title: Low-dose CT-based Method for Detection of Subclinical Anthracycline-induced Cardiotoxicity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Anna Narezkina, Assistant Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 160252
Record Dates: First submitted 2018-01-24; First posted 2018-06-12 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT monitoring arm (Experimental): 18-75 year old patients with newly-diagnosed cancer, scheduled to undergo anthracycline-based chemotherapy.
  Interventions: Diagnostic Test: low dose CT

INTERVENTIONS:
Diagnostic Test: low dose CT — CT-based protocol for detection of anthracycline-induced myocardial dysfunction at early stages

SUMMARY:
Prospective single arm study to evaluate a low-dose CT-based protocol for early detection of myocardial dysfunction in 50 cancer patients undergoing anthracycline-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent.
2. 18-75 year old patients with newly-diagnosed cancer scheduled to undergo anthracycline-based chemotherapy (minimum of 200 mg/m2 of doxorubicin or equivalent) at UCSD Medical Center.
3. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   • A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months)
4. Women of child-bearing potential must have a negative pregnancy test during the screening period.

Exclusion Criteria:

1. Prior chemotherapy with anthracycline;
2. Persistent tachycardia (heart rate>90);
3. LVEF<53% or history of cardiomyopathy or decompensated heart failure;
4. Baseline GLS below lower limit of normal (normal range varies depending on age and gender (23)) or inability to obtain meaningful strain data due to poor quality of Echocardiographic images;
5. Known unrevascularized coronary artery disease, myocardial infarction within 30 days of enrollment;
6. Moderate or severe valvular heart disease;
7. Prior allergy or intolerance to iodinated contrast;
8. Renal failure (GFR<30, creatinine >1.5);
9. Cancer involvement of the heart.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
cardiomyopathy | 12 months after completion of chemotherapy
  Cardiomyopathy is defined as a decrease in the left ventricular ejection fraction by echocardiography of greater than 10 percentage points, to a value < 53% (normal reference value for 2D echocardiography).

SECONDARY OUTCOMES:
Change in CT-based left ventricular strain parameters | 12 months after completion of chemotherapy
  Change in CT-based left ventricular strain parameters before and after the chemotherapy
Change in left ventricular global longitudinal strain based on echocardiography | 12 months after completion of chemotherapy
  Change in left ventricular global longitudinal strain between baseline and post-chemotherapy.
Change in echocardiographic left ventricular ejection fraction | 12 months after completion of chemotherapy
  left ventricular ejection fraction change between baseline and post-chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Narezkina, MD, Principal Investigator — UCSD
Locations (1):
- University of California San Diego Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No